CLINICAL TRIAL: NCT03170635
Title: The Refreshing Recess Program for Promoting Student Participation and Enjoyment: An Outcome Study
Brief Title: Refreshing Recess: Staff and Student Feedback Outcome Study (EMCRR)
Acronym: (EMCRR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Susan Bazyk, Professor, Occupational Therapy, Cleveland State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 29788-BAZ-HS
Record Dates: First submitted 2017-05-19; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Interpersonal Relations; Occupational Therapy
Keywords: recess, occupational therapy

STUDY DESIGN:
Intervention Model Description: The Refreshing Recess program was provided one day/week for 6 consecutive weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 week Refreshing Recess program (Other): Education and coaching for recess supervisors to learn about how to promote positive social interaction and active play with all students during recess. Provision of play activities for students during recess that foster active play, teamwork, and inclusion of students with disabilities and/or social challenges.
  Interventions: Behavioral: Refreshing Recess program

INTERVENTIONS:
Behavioral: Refreshing Recess program — 6-week program integrated into recess in order to build capacity of recess supervisors to foster active play and socialization so that all students enjoy recess and socialization with peers.

SUMMARY:
A mixed methods design was used to explore the outcomes of a 6-week, occupational therapy-led Refreshing Recess program designed to build capacity of recess supervisors to create a positive recess experience so that all students can successfully participate in and enjoy active play and socialization with peers.

DETAILED DESCRIPTION:
A mixed methods design was used to explore the outcomes of a 6-week, occupational therapy-led Refreshing Recess program designed to build capacity of recess supervisors to create a positive mealtime environment so that all students can successfully participate in and enjoy recess and socialization with peers. Occupational therapy practitioners provide weekly information and coaching to recess supervisors and embed weekly activities into the recess experience (e.g. team building games, strategies for including students with disabilities, etc.).

ELIGIBILITY:
Inclusion Criteria:

* all kindergarten through 4th grade students in school where the Refreshing Recess program was offered based on principal approval
* all recess supervisors who supervised recess during program implementation

Exclusion Criteria:

- students who did not receive the school-sponsored Refreshing Recess program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in students' participation and enjoyment of recess play and socialization | pretest prior to the program implementation (10 minutes) and posttest 6 weeks later after program implementation (10 minutes)
  Visual analogue survey

SECONDARY OUTCOMES:
Changes in recess supervisors knowledge, beliefs, and actions related to supervising recess | pre-survey prior to program implementation (10 min.) and post-survey following the 6 week program (10 min.)
  Likert scale survey

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bazyk, Principal Investigator — Cleveland State University

IPD SHARING:
Plan to Share IPD: No